CLINICAL TRIAL: NCT06665178
Title: Whole Genome and Transcriptome Tumor Sequencing to Identify Predictors of Sensitivity to Sequential Sacituzumab Govitecan (SG) Following Trastuzumab Deruxtecan (T-DXd) Treatment in ER+/HER-2 Low Metastatic Breast Cancer
Brief Title: Genomic and Transcriptomic Predictors of Sequential SG Sensitivity After T-DXd in ER+/HER2-Low Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Stephen Chia, Medical Oncologist, BC Cancer, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG6822
Record Dates: First submitted 2024-10-18; First posted 2024-10-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (Experimental): Patients will receive SG at an initial dose of 10 mg per kilogram intravenously on day 1 and 8 of 21 day cycles.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Administer Sacituzumab Govitecan (SG) at 10 mg/kg as an intravenous (IV) infusion on Days 1 and 8 of a 21-day cycle. SG should not be administered as an IV push or bolus.

SUMMARY:
Advanced hormone positive (HR+), HER2 negative breast cancer continues to pose a challenge when patients have progressed on CDK4/6 inhibitor and endocrine therapy leaving limited treatment options. Antibody-drug conjugates (ADCs) such as sacituzumab govitecan (SG) and trastuzumab deruxtecan (T-DXd) have changed practice due to significant improvement in progression free survival (PFS) and overall survival (OS) seen in this disease setting. There is a genuine interest to use SG sequentially after T-DXd, however there is no current prospectively curated evidence to support this strategy. Though the epitope is different, the payload are both topoisomerase I inhibitors. Thus, evidence is needed of both clinical efficacy and identification of mechanisms of sensitivity and resistance to sequential ADCs in HER-2 low MBC.

It is hypothesized that performing whole genome and whole transcriptome sequencing in fresh tumour biopsies post progression of T-DXd and prior to SG in ER+/HER2 low metastatic breast cancer (MBC) will provide mechanistic insights into identifying biomarkers, and thus patients, sensitive to sequential SG.

DETAILED DESCRIPTION:
This is a prospective single-centre Canadian study (BC Cancer Vancouver) enrolling ER+/HER2 low MBC with disease progression after at least one line of endocrine therapy in combination with a CDK 4/6 inhibitor and at least one line of chemotherapy which must include T-DXd as the immediate prior line of treatment in the advanced stage setting.

Patients will receive SG at an initial dose of 10 mg per kilogram intravenously on day 1 and 8 of 21 day cycles. Treatment will continue until evidence of progressive disease, significant toxicity in which patient and or physician wishes to discontinue treatment and/or patient or physician desire to discontinue treatment for any reason.

Tumor specimens will collected from biopsies between the time of informed consent and prior to first administration of SG. The pathology will be reviewed and nucleic acids extracted. Constitutional DNA representing normal cells will be extracted from peripheral blood. PCR-free DNA libraries and either strand-specific or ribo-depleted RNA libraries will be constructed. Following which whole genome sequencing and transcriptome sequencing will be performed.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Willing and able to provide signed informed consent approved by UBC/BC Cancer REB
2. Female or male patients, regardless of race and ethnic group, who are ≥18 years old at the time of informed consent
3. Patients with locally advanced or metastatic ER+/HER2 low (defined as IHC 1+ or 2+ but FISH or CISH negative by ratio as per ASCO/CAP guidelines) breast cancer. Patients with imaging confirmed inoperable locally advanced breast cancer for which treatment is palliative in intent are also permitted.
4. Prior treatment must have included prior endocrine based treatment in the metastatic setting in conjunction with a CDK4/6 inhibitor.
5. Prior treatment must include at least 1 line of chemotherapy which must include trastuzumab deruxtecan (T-DXd) as the immediate prior line of therapy prior to study enrollment
6. The tumour must be accessible to be able to safely perform image guided biopsies for WGS and WTS.
7. Negative serum pregnancy test at baseline for pre-menopausal patients (within 14 days prior to randomization) and agreement to use medically approved precautions to prevent pregnancy during the study and for 12 weeks following the last dose of SG
8. Patients can have measurable or non measurable (but assessable) disease by CT or MRI as per RECIST Version 1.1 criteria as evaluated locally. Tumor lesions situated in a previously irradiated area are considered measurable if unequivocal progression has been documented in such lesions since radiation.
9. ECOG PS 0-2
10. Life expectancy ≥ 3 months
11. Acceptable bone marrow and organ function defined by the following laboratory values:

    1. Absolute neutrophil count ≥1.0 x 109/L
    2. Platelets ≥100 x 109/L
    3. Hemoglobin ≥9.0 g/dL
    4. INR ≤1.5
    5. Serum creatinine clearance >50 mL/min
    6. In absence of liver metastases, direct bilirubin ≤1.5 x ULN, ALT and AST should be below ≤2.5 x ULN. If the patient has liver metastases, ALT and AST should be < 5.0 x ULN.
12. Controlled brain metastasis (as per clinical determination) is allowed in the study at least 4 weeks before treatment. (Controlled brain metastasis is defined as no longer symptomatic from brain metastasis or no longer requiring higher doses of corticosteroids (> 10 mg Dexamethasone per day) for CNS management. Anticonvulsants and stable corticosteroids dose can be included in the study).

Exclusion Criteria

Patients who meet any of the following exclusion criteria are not eligible to be enrolled in this study:

1. Patient is currently participating in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Patient has a known hypersensitivity to SG, irinotecan or its active metabolite SN-38.
3. Patients not available for follow up
4. Patients who are not willing to consider systemic treatment options
5. Tumor not accessible or not safe to perform biopsies
6. Patient has not had resolution of all acute toxic effects of prior anti-cancer therapy to CTCAE v. 5.0 grade ≤1 (except toxicities not considered a safety risk for the patient at investigators discretion: e.g. grade 2 peripheral neuropathy from prior chemotherapy that is stable).
7. Have an active second malignancy. Patients with a history of malignancy that has been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (e.g. non-melanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
8. Have known active central nervous system (CNS) metastases. Patients with previously treated brain metastases may participate provided they have stable CNS disease (defined as no longer symptomatic from brain metastasis or no longer requires higher doses of corticosteroids (> 10 mg Dexamethasone per day) for CNS symptom management. Anticonvulsants and stable corticosteroids dose can be included in the study). Screening for brain metastasis not required for enrollment.
9. Pregnancy and breast feeding
10. Patient without an adequate hematologic, renal and hepatic function as per above inclusion criteria
11. Patient has a pre-existing condition with uncontrolled diarrhea, chronic inflammatory bowel disease or GI perforation within 6 months prior to enrollment.
12. Have active serious infection requiring antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Altered Tumor Genes by PFS Duration on SG Post T-DXd | Up to an average of 6 months
  Number and identification of altered/mutated genes in the tumors in the subgroup of patients with a longer PFS on SG post T-DXd compared to the tumors in the subgroup of patients with a shorter PFS on SG post T-DXd.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to an average of 6 months
  Progression free survival (PFS) of SG post T-DXd in ER+/HER2 low MBC as measured by RECIST criteria
Response rate (RR) | Up to an average of 6 months
  Response rate (RR) of SG post T-DXd as measured by RECIST 1.1 criteria
Grade 2-4 toxicities | Up to an average of 3 months
  Number of Participants with the CTCAE version 5 grade 2-4 toxicities reported in SG post T-DXd in ER+/HER2 low MBC
Overall survival | Up to an average of 12 months
  Overall survival of SG post T-DXd
Trop-2 expression and HER-2 expression | Up to an average of 12 months
  Trop-2 expression and HER-2 expression by IHC in the metastatic biopsy and correlation with PFS and RR
Dose intensity | Up to an average of 3 months
  Dose intensity (with and without growth factor support) of SG delivered post T-DXd in ER+/HER2 low MBC

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modi S, Jacot W, Yamashita T, Sohn J, Vidal M, Tokunaga E, Tsurutani J, Ueno NT, Prat A, Chae YS, Lee KS, Niikura N, Park YH, Xu B, Wang X, Gil-Gil M, Li W, Pierga JY, Im SA, Moore HCF, Rugo HS, Yerushalmi R, Zagouri F, Gombos A, Kim SB, Liu Q, Luo T, Saura C, Schmid P, Sun T, Gambhire D, Yung L, Wang Y, Singh J, Vitazka P, Meinhardt G, Harbeck N, Cameron DA; DESTINY-Breast04 Trial Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Low Advanced Breast Cancer. N Engl J Med. 2022 Jul 7;387(1):9-20. doi: 10.1056/NEJMoa2203690. Epub 2022 Jun 5. PMID 35665782
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- See also: Jones, S.J., Laskin, J., Li, Y.Y. et al. Evolution of an adenocarcinoma in response to selection by targeted kinase inhibitors. Genome Biol 11, R82 (2010). — https://doi.org/10.1186/gb-2010-11-8-r82
- See also: Pleasance E, Titmuss E, Williamson L et al. Pan-cancer analysis of advanced patient tumors reveals interactions between therapy and genomic landscapes. — https://www.nature.com/articles/s43018-020-0050-6